CLINICAL TRIAL: NCT06070766
Title: Can Digital Health Technology Guide Medical Providers, in Treating Chronic Conditions With RIVER Ketamine Protocols Safely at Home?
Brief Title: RIVER At Home Ketamine Protocols
Status: Recruiting | Type: Observational
Sponsor: RIVER Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: RIVER IRB IRB00013708 2023-2
Record Dates: First submitted 2023-09-22; First posted 2023-10-06 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Chronic Condition; Chronic Pain; Chronic Disease; Major Depressive Disorder; Post Traumatic Stress Disorder; Anxiety Disorders
Keywords: Ketamine; Neuroinflammation; Auricular
MeSH Terms: conditions — Chronic Disease; Chronic Pain; Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Anxiety Disorders; Neuroinflammatory Diseases | interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (13):
- Chronic Pain: Drug: Ketamine The efficacy of the various approaches to prescribing Ketamine currently in use off-label. The focus will be to include ketamine research within the treatment plan of those with chronic conditions. A RIVER Ketamine protocol will be developed
  Interventions: Drug: Ketamine
- Anxiety: Drug: Ketamine The efficacy of the various approaches to prescribing Ketamine currently in use off-label. The focus will be to include ketamine research within the treatment plan of those with chronic conditions. A RIVER Ketamine protocol will be developed
  Interventions: Drug: Ketamine
- Veterans and First Responders: The efficacy of the various approaches to prescribing Ketamine currently in use off-label. The focus will be to include ketamine research within the treatment plan of those with chronic conditions. A RIVER Ketamine protocol will be developed
  Interventions: Drug: Ketamine
- Depression: Drug: Ketamine The efficacy of the various approaches to prescribing Ketamine currently in use off-label. The focus will be to include ketamine research within the treatment plan of those with chronic conditions. A RIVER Ketamine protocol will be developed
  Interventions: Drug: Ketamine
- Trauma: Drug: Ketamine The efficacy of the various approaches to prescribing Ketamine currently in use off-label. The focus will be to include ketamine research within the treatment plan of those with chronic conditions. A RIVER Ketamine protocol will be developed
  Interventions: Drug: Ketamine
- Auricular Chronic Pain: Auricular Therapy (Ear acupuncture)
  1. National Acupuncture Detoxification Association
  2. Battlefield Acupuncture
  Interventions: Drug: Ketamine
- Auricular Anxiety: Auricular Therapy (Ear acupuncture)
  1. National Acupuncture Detoxification Association
  2. Battlefield Acupuncture
  Interventions: Drug: Ketamine
- Auricular Depression: Auricular Therapy (Ear acupuncture)
  1. National Acupuncture Detoxification Association
  2. Battlefield Acupuncture
  Interventions: Drug: Ketamine
- Auricular Trauma: Auricular Therapy (Ear acupuncture)
  1. National Acupuncture Detoxification Association
  2. Battlefield Acupuncture
  Interventions: Drug: Ketamine
- Chronic Pain MH: 4. Millennium Health The Phase 2 Protocol (P2P) has entered its 4th year of application in those with symptoms associated with all forms of traumatic brain injury (T.B.I.). Listening to any of the following Joe Rogan Experience podcasts, 1589, 1056, or 700, will provide a number of discussions on this topic. Since the 2020 pilot study with active duty Marines (U.S.M.C.), looking at the benefits of a 100% nutraceutical approach to T.B.I., precipitated changes in mental and physical health, we had the start to developing the P2P. With over 8,000 participants, we see the benefits derived from the 2023 Phase 2 Protocol.
  Interventions: Drug: Ketamine
- Anxiety MH: 4. Millennium Health The Phase 2 Protocol (P2P) has entered its 4th year of application in those with symptoms associated with all forms of traumatic brain injury (T.B.I.). Listening to any of the following Joe Rogan Experience podcasts, 1589, 1056, or 700, will provide a number of discussions on this topic. Since the 2020 pilot study with active duty Marines (U.S.M.C.), looking at the benefits of a 100% nutraceutical approach to T.B.I., precipitated changes in mental and physical health, we had the start to developing the P2P. With over 8,000 participants, we see the benefits derived from the 2023 Phase 2 Protocol.
  Interventions: Drug: Ketamine
- Depression MH: 4. Millennium Health The Phase 2 Protocol (P2P) has entered its 4th year of application in those with symptoms associated with all forms of traumatic brain injury (T.B.I.). Listening to any of the following Joe Rogan Experience podcasts, 1589, 1056, or 700, will provide a number of discussions on this topic. Since the 2020 pilot study with active duty Marines (U.S.M.C.), looking at the benefits of a 100% nutraceutical approach to T.B.I., precipitated changes in mental and physical health, we had the start to developing the P2P. With over 8,000 participants, we see the benefits derived from the 2023 Phase 2 Protocol.
  Interventions: Drug: Ketamine
- Tramua MH: 4. Millennium Health The Phase 2 Protocol (P2P) has entered its 4th year of application in those with symptoms associated with all forms of traumatic brain injury (T.B.I.). Listening to any of the following Joe Rogan Experience podcasts, 1589, 1056, or 700, will provide a number of discussions on this topic. Since the 2020 pilot study with active duty Marines (U.S.M.C.), looking at the benefits of a 100% nutraceutical approach to T.B.I., precipitated changes in mental and physical health, we had the start to developing the P2P. With over 8,000 participants, we see the benefits derived from the 2023 Phase 2 Protocol.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — The use of ketamine in chronic conditions.
  Other Names: Ketalar

SUMMARY:
Multiple site studies with the recruitment of other sub-investigators and sites. It's sobering to consider how chronic illness makes us more vulnerable to suicidal thoughts and behavior. However, the existence of multiple risk factors also means that there are numerous ways to intervene. Addressing and improving even one risk area will reverberate and improve other areas and the quality of life.

RIVER Foundation is completing a 500-participant pilot study researching the safety of oral and nasal ketamine at home with no therapy. The pilot study examined three psychological scales: P.H.Q. 9, G.A.D. 7, and PCL5 scores. The interim report will be available in Nov 2023 with a final report in June 2024.

The lack of knowledge for the average medical practitioner makes ketamine a boutique medicine, often costly and unaffordable to those in need. Yet daily medical providers are eliminating ketamine as a choice in the treatment of chronic conditions.

The pilot study demonstrated the who, and where. The who, was adults with a chronic condition. The pilot study demonstrated the majority of those who could use ketamine are not receiving it due to cost. According to the 500-participant study, ketamine is safe and effective for at-home use thus demonstrating the where (at home with no supervision).

DETAILED DESCRIPTION:
The why, when, what, and how much needs to be studied. The new study is five years and up to 50,000 participants. With digital technology, many questions can be answered. The study is a pay-to-participate study in which minimal fees will be charged for the technology.

Lacking in the original RIVER pilot study was when and how often the participants would take their medication (Ketamine) and which additional add-on protocols make the treatments more effective. The RIVER protocol was not based on weight but on the severity of symptoms, history of chronic conditions, and current medications.

Adverse effects were standard nausea; however, there were only three minor adverse effects. None of the effects were severe enough to halt the research. The results were promising. Drops in PHQ9 depression scores were reduced overall between 25% and 61%. RIVER Ketamine protocols were developed, making home use safe and effective.

Suicide rates increased approximately 36% between 2000-2021. Suicide was responsible for 48,183 deaths in 2021, about one every 11 minutes. The number of people who think about or attempt suicide is even higher. In 2021, an estimated 12.3 million American adults seriously thought about suicide, 3.5 million planned a suicide attempt, and 1.7 million attempted suicides.

Oral Ketamine offers a promising pharmacologic adjunct to chronic condition treatments. It may offer a more approachable alternative to IV or I.M. Ketamine. The results of the RIVER pilot study warrant further investigation into the safety and efficacy of oral Ketamine for chronic conditions.

Oral Ketamine is only available at a compounding pharmacy, which can lead to fluctuations in dosing. Oral Ketamine is used off-label and is becoming a front-line medicine in treating chronic conditions. Dosing becomes an issue with using multiple compounding pharmacies. In the pilot study, River Foundation contracted with one pharmacy, Precision Compounding Pharmacy. RIVER Foundation received accurate dosing and documentation.

Psychedelic therapies involving Ketamine have gained considerable attention for their potential to facilitate transformative experiences and promote mental well-being. Ketamine is being explored to treat various mental health conditions, such as post-traumatic stress disorder, depression, and substance abuse.

The U.S. population suffers from chronic conditions that impact a person's daily living. (45% in 2018; Raghupathi & Raghupathi). Individuals suffering from a chronic condition are three times more likely to complete suicide, leading to approximately 800,000 people dying by suicide each year worldwide. Additionally, nonfatal self-injurious behavior occurs 20x more frequently.

"From 2006 to 2013, aggregate E.D. plus inpatient costs of E.D. visits related to suicidal idealization that resulted in admission to the same hospital increased from $600 million to $2.2 billion-an average annual increase of 20.4 percent. Aggregate costs of these E.D. visits rose faster than the actual number of visits, which increased by only 16.2 percent on average annually from 2006 to 2013."

"Depression is one of the most common mental disorders and can cause tremendous challenge and burden for individuals and families. It also carries a large economic cost. The economic burden of major depressive disorder among U.S. adults was an estimated $236 billion in 2018, an increase of more than 35% since 2010 (year 2020 values), according to research published in early May in the journal Pharmacoeconomics.

The increase has been greater among younger adults. Young adults, 18 to 34 years, accounted for nearly half (48%) of adults with depression in 2018, up from 35% in 2010. Young adults have also been especially impacted by the COVID-19 pandemic. Throughout the pandemic, young adults have experienced higher levels of depression and anxiety compared to older adults. An estimated 36% of 18-29-year-olds were experiencing symptoms of depression in early May 2021, compared to 22% of those 40-49 and 15% of those age 50-59, according to the Centers for Disease Control and Prevention's (C.D.C.) Household Pulse Survey."

Research is up-and-coming on the use of Ketamine. One study out of the University of Alabama found great success with Ketamine and suicidal ideation (S.I.).

"We found Ketamine to alleviate suicidal ideation at 90, 120, and 180 min after infusion according to the B.S.S. and at 120 min according to the MADRS-SI score. Remission from suicidal ideation was defined by a score of 2 or less on the MADRS-SI item (indicating fleeting suicidal thoughts or less). Ninety minutes after infusion, eight of nine subjects of the ketamine group had remission (88%) compared with three of nine (33%) in the placebo group (p < .05

…The change in depression is a secondary outcome. The reduction in depression fell just short of a statistically significant difference. This reduction was rapid with the nadir effect three days after infusion."

Depressed patients often present to the emergency department with complaints of suicidal thoughts, which accounts for more than half a million admissions annually to the emergency department in the United States.

Suicide is the 10th leading cause of death in the United States (Heron, 2016), and suicide rates are rising alarmingly. With the recent lockdowns of COVID, the increase is even more rapid.

"In the absence of specific treatments for acute S.I., most suicidal patients are hospitalized for brief stabilization and are often discharged before psychopharmacological treatments can show efficacy. No strong evidence exists to demonstrate that brief inpatient hospitalizations are associated with a significant reduction in suicidal potential. Thus, there is an urgent need to pursue treatment options for suicidal ideation, especially in emergency department settings." Ketamine is being described as the next wonder drug in psychiatry. Psychiatric disorders have a limited number of treatments approved by the F.D.A. With the lack of FDA-approved prescription medicine, the highest rates of off-label prescriptions are for psychotropic medications.

Off-label prescribing with limited proof of efficacy is commonplace with psychotropic medications. In recent studies in community clinical practices, 40 to 80 percent of recipients of commonly prescribed psychotropic medications (including antidepressants, antipsychotics, and anticonvulsants) were receiving these medications for off-label indications.

In the primary care setting, a survey on antidepressant medications showed that 84.2 percent of off-label prescriptions had no convincing evidence of efficacy for the indication. Off-label prescription has consistently presented a significantly increased risk of adverse drug events in different patient populations.

The data shows that Ketamine could significantly save billions of dollars annually. As with any generic drug, there is no incentive to spend millions of dollars to go through the F.D.A. process of relabeling when it is legal to use as is.

Commercially available Ketamine comes in three variants: R/S, S, and R. An unexpected finding was the ability of racemate ketamine as a rapid onset and sustained antidepressant for patients with treatment-resistant depression. Racemate (R) Ketamine is Schedule III and is not FDA-approved for treating any psychiatric disorder. The use of R Ketamine for any use other than as an anesthetic is classified as off-label.

However, the "S" form of Ketamine, which is derived from Ketamine and known as Spravato (esketamine), is a Schedule III controlled substance that was approved by F.D.A. in 2019 as a nasal spray for treatment-resistant depression in adults and depressive symptoms in adults with major depressive disorder with acute suicidal ideation or behavior, in conjunction with an oral antidepressant.

The ketamine molecule contains an asymmetrical carbon atom with two enantiomers. The S (+) isomer is three times more potent and longer acting than the R (-) isomer.

Ketamine contains a chiral center at the C-2 carbon of the cyclohexanone ring so that two enantiomers exist, S (+) ketamine and R (-) ketamine. Commercially available racemic ketamine preparations (such as Ketalar) contain equal concentrations of the two enantiomers. The dextro-S(-)-isomer of Ketamine has approximately 3- to 4-fold the potency of the levo-R(-)- isomer.85 The S(+)-isomer appears to be cleared more rapidly than the R(-) isomer, resulting in a shorter duration of effect and more rapid recovery. (Adams et al., 1994)

Equipotent doses of the S(+)-isomer and the racemate appear to have similar effects on physiologic parameters. Evidence suggests that the R(-)-isomer produces a higher rate of emergence reactions and more agitated behavior than the S(+) isomer. (Geisslinger et al., 1999) It has been known since the late 1970s that the ketamine enantiomers exhibit pharmacologic and clinical differences. Receptor studies in animal models show that S(+) ketamine has approximately fourfold greater affinity at phencyclidine binding sites on the NMDA receptor than R(-) Ketamine.

Not all of Ketamine's effects are stereoselective. Norepinephrine release is inhibited in a nonstereoselective manner at clinically relevant concentrations. However, its uptake is influenced stereoselectively: both isomers inhibit neuronal uptake, whereas S(+) ketamine additionally inhibits extraneuronal uptake. Muscarinic receptors and Ca channels are inhibited nonstereoselectively. Interestingly, serotonin transport is inhibited twofold more potently by R(-) Ketamine. (Schwartzman et al 2011)

Animal studies have not revealed significant pharmacokinetic differences between the enantiomers and the racemic mixture. After subcutaneous application, similar plasma and brain concentration curves have been found. In a clinical study, however, a significantly higher elimination rate was observed for S(+) Ketamine compared with the racemate.

The increased inhibitory potency at the NMDA receptor combined with similar pharmacokinetics suggests that S(+) ketamine may be an interesting clinical drug, and its pharmacological properties have been studied in some detail.

Recent research suggests that neuroinflammation, an immune response in the brain, may have counter-productive effects on the efficacy of these psychedelic treatments. Vital to the ability of Ketamine to affect a change in neuronal functioning that leads ultimately to improved mental health is the ability to be recognized by specific cell receptors.

In the presence of neuroinflammation, most frequently induced by trauma, is a change in the composition of the brain's biochemistry from one that is neuro-permissive to that of neuro-restrictive.

Neurons and glial cells exposed to a neuropermissive environment function optimally, producing neurotransmitters, enzymes, neuroreceptors, neurosteroids, and various neurochemicals to support a healthy brain. Contrary to this is a neurorestrictive environment that induces activation of glial cells with the release of pro-inflammatory cytokine that fosters an increase in oxidative stress, leading to more inflammation, mitochondrial dysfunction, apoptosis, and loss of neurotransmitters and their receptors.

It's important to note that the effects of psychedelic medications on brain function are complex and can vary depending on the individual, the dose, and the composition of the brain's neurochemistry. This paper is not about delivering Ketamine but optimizing its beneficial effects by modifying and controlling adverse conditions such as neuroinflammation.

Think of neuroinflammation as a wall that needs to be surmounted by the psychedelic agent. Lowering this barrier will allow for micro-dosing efficacy to be enhanced, as well as improving the surrounding neurochemistry to support the biological changes induced by the Ketamine.

ELIGIBILITY:
Inclusion Criteria:

Must have an identifiable chronic condition.

Exclusion Criteria:

Healthy Population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with chronic conditions need either their mental health or pain controlled.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Mental Health PHQ9 | Through study completion, an average of 5 years
  The use of psychological scales to measure participants' mental health with the use of ketamine.
  The Patient Health Questionnaire-9 (PHQ9), Patient Health Questionnaire 9 has a possible range of 0-27. Zero being no depression and 27 being severe depression. A multiline graph will show the results of PHQ9 will be produced.
Mental Health GAD7 | Through study completion, an average of 5 years
  Participants will be screened using the Generalized Anxiety Disorder-7 (GAD7) with a total score for the seven items ranging from 0 to 21. Scores 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety, respectively.
  Participants will be given a baseline survey and will be given a survey to complete throughout the study. A multiline graph will show the results of the GAD7 will be produced.
Mental Health PCL5 | Through study completion, an average of 5 years
  Participants will be screened using the Posttraumatic Stress Disorder Checklist (PCL-5) PCL-5. On a 4-point scale, scores can be tabulated for individual items to give information about the severity of the four DSM-5 symptom clusters. If a score of 2 (moderate) is considered to be a positive endorsement of a given criterion, the PCL-5 can be used in combination with a clinical interview to make a provisional DSM-5 diagnosis. Testing the PCL-5 with veterans has determined a score of 31 to 33 to be a valid cutoff for a positive screen. The scores range from 0-80, 0 being no symptoms to extreme issues with post-traumatic stress disorder. A multiline graph will show the results of the amount of ketamine and the PCL5 will be produced.

SECONDARY OUTCOMES:
Auricular Therapy | Through study completion, an average of 5 years
  Participants using auricular therapy will be documented and a separate graph will be produced for each month's use of auricular therapy during the study. The graph will document only if the articular therapy is used.
Millennium Health | Through study completion, an average of 5 years
  Since the 2020 pilot study with active duty Marines (U.S.M.C.), looking at the benefits of a 100% nutraceutical approach to T.B.I., precipitated changes in mental and physical health, we had the start to developing the P2P. A graph will be produced to demonstrate each month of the use of Millennium Health.

CONTACTS AND LOCATIONS:
Overall Officials: Dharma Rose, D.O. M.S., Principal Investigator — RIVER Foundation; Frank Yurseak, Ph.D., Study Chair — RIVER Foundation; Jeffery Newton, Principal Investigator — RIVER Foundation; Alejandro Fernandez, Principal Investigator — RIVER Foundation; James Taggart, MD, Principal Investigator — RIVER Foundation; Ed Lesofski, MS, Study Director — RIVER Foundation
Locations (2):
- United States (2):
  - RIVER Foundation, Bigfork, Montana
  - RIVER Telehealth, Helena, Montana